CLINICAL TRIAL: NCT06122558
Title: Efficacy of Probiotic in Patients With Functional Constipation
Brief Title: Efficacy of Probiotic Against Functional Constipation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Tze LIONG (Other)
Collaborators: Deyang People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Min-Tze LIONG, Professor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DCPH-2023-03-001-K01; P-ID0024/21(R) (Other: Universiti Sains Malaysia)
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Constipation - Functional
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Probiotic Lactobacillus plantarum at 9 log CFU/day for 8 weeks
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g of maltodextrin, administered daily for 8-weeks)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic Lactobacillus plantarum at 9 log CFU/day for 8 weeks
  Arms: Probiotic
Dietary Supplement: Placebo — Intervention consists of daily administration of 2g of maltodextrin, administered daily for 8-weeks)
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotic in modulating gut microbiota and treating functional constipation in patients aged 18-81.

DETAILED DESCRIPTION:
Constipation is a common clinical intestinal functional disease worldwide, and its main manifestations are difficulty in defecation and/or decreased frequency of defecation. Difficulty defecating includes straining, difficulty passing, sensation of incomplete defecation, sensation of anorectal blockage, time-consuming defecation, and need for assistance, fewer bowel movements are fewer than 3 bowel movements per week and the duration of chronic constipation is at least 6 months.

The quality of life of patients with chronic constipation is significantly lower than that of non-chronic constipation patients. Some patients have a heavy financial burden due to abuse of laxatives or repeated visits to doctors, including visits to doctors, examinations, direct economic losses caused by treatment and hospitalization and indirect economic losses caused by reduced work productivity and absenteeism.

Constipation caused by functional diseases is mainly caused by nerve smooth muscle dysfunction in the colon, rectum and anus, including functional constipation, functional defecation disorder and constipation-predominant irritable bowel syndrome. In some cases, functional constipation may be related to normal or slow colonic transit and/or bowel dysfunction (pelvic floor dysfunction).

Constipation treatment methods include basic treatment measures such as increasing dietary fiber and water, increasing exercise and other lifestyles, and establishing good bowel habits. Volumetric laxatives and osmotic laxatives are options for patients with mild to moderate constipation. Stimulant laxatives may be used as a short-term/intermittent remedy.

In recent years, the treatment of chronic constipation patients with probiotics has been proposed. Existing research data confirm that patients with chronic constipation have intestinal microecological imbalance. Studies have shown that Bifidobacterium, Lactobacillus, dominant bacterial groups such as Bacteroides decreased significantly, while Escherichia coli, Staphylococcus aureus, Enterobacteriaceae (Citrobacter, Klebsiella, etc.) and fungi and other potential pathogenic bacteria increased significantly, and this trend was related to the severity of constipation. Although probiotics are not the first-line drugs for the treatment of chronic constipation, they can promote intestinal peristalsis and restoration of gastrointestinal motility. Possible mechanisms include changes in the number and types of intestinal flora; metabolites of the flora (methane and short-chain fatty acids), cellular components of bacteria (lipopolysaccharides) or the interaction between bacteria and the host immune system affects a variety of gut functions. Gut microbes through the digestion of polysaccharides in the gut produce short chain fatty acids (short chain fatty acids, SCFAs) to provide energy for the body. SCFAs produced by intestinal flora metabolism also inhibits the growth of pathogenic bacteria and reduces the accumulation of phenolic substances produced by pathogenic bacteria, promote intestinal peristalsis to relieve constipation symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for functional constipation in the Rome IV
* Ruled out for IBS or secondary constipation

Exclusion Criteria:

* Diagnosed with refractory constipation
* Any other constipation caused by neurological diseases, metabolic diseases, obstructive diseases and drugs
* Mental illness
* Immunodeficiency diseases or used immunosuppressants, serious diseases of the heart, brain, kidney and other systems, malignant tumors, intestinal perforation, intestinal obstruction, intestinal bleeding
* Currently using antibiotics or have a history of taking antibiotics in the past 4 weeks.
* Participating in other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in patients with functional constipation upon administration of probiotic or placebo | 8-weeks
  Differences in microbiota abundance in fecal sample of patients with functional constipation upon administration of probiotic compared to placebo as assessed via DNA profiling of fecal samples upon Ilumina MiSeq sequencing

SECONDARY OUTCOMES:
Constipation profiles of patients with functional constipation upon administration of probiotic or placebo | 8-weeks
  Differences in constipation profiles in patients with functional constipation upon administration of probiotic compared to placebo as assessed via number of complete spontaneous bowel movement (CSBM) per week and bowel habits
Quality of life profiles of patients with functional constipation upon administration of probiotic or placebo | 8-weeks
  Differences in QoL profiles in patients with functional constipation upon administration of probiotic compared to placebo as assessed via the Hamilton Anxiety Scale (HAM-A) comprising of 14-items, with a 5-point Likert scale (8-56 points), where a higher score indicates more severe anxiety symptoms
Defecation profiles of patients with functional constipation upon administration of probiotic or placebo | 8-weeks
  Differences in defecation profiles in patients with functional constipation upon administration of probiotic compared to placebo as assessed via the balloon expulsion test (time to expel the balloon)
Defecation profiles of patients with functional constipation upon administration of probiotic or placebo | 8-weeks
  Differences in defecation profiles in patients with functional constipation upon administration of probiotic compared to placebo as assessed via pelvic floor muscle electromyography
Immunity profiles of patients with functional constipation upon administration of probiotic as assessed via blood samples | 8-weeks
  Differences in concentrations of proteins such as interleukins (IL-10, IL-4, IL-6, Tumour Necrosis Factor-alpha, Interferon gamma) in blood samples of patients upon administration of probiotic compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Min Liong, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (2):
- Deyang People's Hospital, Deyang, Sichuan, China
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No